CLINICAL TRIAL: NCT03320109
Title: Vitamin D Status and Intakes and Their Association With Cognitive Trajectory in a Longitudinal Study of Urban Adults
Brief Title: Serum, Dietary and Supplemental Vitamin D's Association With Cognitive Decline
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, May Ahmad Baydoun, Staff Scientist, National Institute on Aging (NIA)
Other Study IDs: NIA2
Record Dates: First submitted 2017-10-20; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Cognitive Decline; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Vitamin D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Vitamin D
  Other Names: Serum 25(OH)D status and dietarysupplemental vitamin D

SUMMARY:
Serum 25(OH)D, dietary and supplemental vitamin D were shown to influence cognitive outcomes in large epidemiological studies. Sex/age-specific and race-specific associations of vitamin D status and intake were examined with longitudinal change in various cognitive domains in a large sample of ethnically and socio-economically diverse US urban adults. Two prospective waves of data from Healthy Aging in Neighborhoods of Diversity across the Life Span (HANDLS) study were used, specifically visit 1: 2004-2009 and visit 2: 2009-2013, mean follow-up time±SD: 4.64±0.93y. Cognitive performance was assessed using 11 test scores covering domains of global cognition, attention, learning/memory, executive function, visuo-spatial/visuo-construction ability, psychomotor speed and language/verbal. Serum 25(OH)D, vitamin D intake and use of supplements containing vitamin D were the key exposures. Multiple mixed-effects linear regression models were conducted, (N=1,231-1,803, k=1.5-2.0 observation/participant).

DETAILED DESCRIPTION:
INTRODUCTION Cognitive impairment, a principal cause for functional disability among the elderly, can lead to dementing illness over time mainly in the forms of Alzheimer's Disease (AD) and vascular dementia (VaD). In fact, AD prevalence is expected to rise, reaching 100 million worldwide by 2050, with 1 in 85 persons potentially living with AD.(1) Thus, uncovering modifiable risk factors that would prevent or delay cognitive impairment is important.

The neuroprotective effects of antioxidant nutrients (e.g. vitamins E) and B-vitamins (e.g. folate) have been at the forefront of cognitive aging and nutritional epidemiology research over the past two decades.(2) Vitamin D's role in preserving cognitive function with aging has recently gained attention in epidemiological investigations.(3) Its public health significance lies in the fact that vitamin D deficiency [25-hydroxyvitamin D3 (25(OH)D)<11 ng/ml (<27.5 nmol/L)] is a highly prevalent condition, particularly among the poor and among African-Americans.(4, 5) Vitamin D is a steroid hormone with its primary function being to regulate body levels of calcium, phosphorus and bone mineralization. While sunlight exposure is its primary source through skin synthesis from 7-dehydrocholesterol, dietary and supplemental intakes of vitamin D play a key role in its overall status. (3) The active form of vitamin D3, namely 1,25-dihydroxy vitamin D3 influences many metabolic pathways through genomic and nongenomic actions which help maintain and stabilize intracellular signaling pathways involved in memory and cognitive function.. (3, 6, 7) The neuroprotective role of vitamin D may be mediated through vasculo-protection and preservation of neurons partly through the expression of neurotrophins and other neurotransmitters which help protect against cognitive dysfunction, through the suppression of inflammatory cytokines.(3, 5, 8) Vitamin D can also down-regulate receptors in memory-relevant regions and enhance amyloid phagocytosis and clearance. (8) Serum 25(OH)D and dietary vitamin D were shown to influence cognitive outcomes in large epidemiological studies. (9-34) This study will examine associations between vitamin D status and intake with longitudinal change in various domains of cognition among a large sample of ethnically and socio-economically diverse US urban adults. It also explores those associations systematically across sex/age groups and race. We hypothesize that both vitamin D status and intake are associated with slower decline in domain-specific cognitive performance over time, but perhaps differentially by age/sex and race.

MATERIALS AND METHODS Database The Healthy Aging in Neighborhoods of Diversity across the Life Span (HANDLS) study is a prospective cohort study initiated in 2004 that focused on the cardiovascular and cognitive health of an ethnically and socio-economically diverse urban population. Specifically, it used area probability sampling to recruit a socioeconomically diverse sample of African American and White urban adults (30-64 years old) residing in thirteen neighborhoods of Baltimore, Maryland.(35) Written informed consent was obtained from participants who were also provided with a protocol booklet and a video that explains study procedures. The study protocol was approved by the National Institute on Environmental Health Sciences Institutional Review Board of the National Institutes of Health. Data for the present study were derived from baseline visit 1 (2004-2009) and the first follow-up examination (visit 2; 2009-2013). Follow-up time ranged from <1y to ~8y, with a mean of 4.64±0.93y.

Study sample HANDLS initially recruited 3,720 participants (Phase I, visit 1). Given that only Phase II had in-depth data including biochemical indices and cognitive performance measures, 25(OH)D was available for 1,981 participants at baseline. The corresponding sample size for dietary and supplemental vitamin D were N=2,177 and N=2,159, respectively. Complete and reliable cognitive tests at each visit varied in sample size as well. Further, the final analytic sample was determined based on exposure and covariate non-missingness at baseline and outcome non-missingness at either visit. Figure 1 describes sample selection for all exposures. The final analytic sizes ranged between N=1,231 and N=1,803 with k=1.5-1.9 observation/participant.

Cognitive assessment Cognitive performance was assessed with 7 tests yielding 11 test scores and covering 7 domains (Global, attention, learning/memory, executive function, visuo-spatial/visuo-construction ability, psychomotor speed, language/verbal): the Mini-Mental State Examination (MMSE), the California Verbal Learning Test (CVLT) immediate (List A) and Delayed Free Recall (DFR), Digit Span Forward and Backwards tests (DS-F and DS-B), the Benton Visual Retention Test (BVRT), Animal Fluency test (AF), Brief Test of Attention (BTA), Trails A and B and the Clock Drawing Test (CDT) (Supplemental method 1). All participants were judged capable of informed consent and were probed for their understanding of the protocol. Although no formal dementia diagnosis was conducted, all participants were given mental status tests, which they completed successfully. In every case, low mental status performance was due to low literacy level without any sign of dementia.

Vitamin D status Total 25(OH)D (in ng/ml) was measured using immunoassay at baseline and follow-up visits. The collected sample was ~0.8 ml of preferably fasting serum which was refrigerated and transported to the lab for analysis. Visit 1 analyses were conducted at the Massachusetts General Hospital.(36) Visit 2 analyses were conducted by Quest Diagnostics, Chantilly, VA.

Dietary vitamin D Dietary factors included in our analyses were measured at the baseline visit. Baseline 24-hour dietary recalls were obtained using the US Department of Agriculture (USDA) Automated Multiple Pass Method, a computerized structured interview.(37) Measurement aids used included measuring cups, spoons, ruler and an illustrated Food Model Booklet. Two recalls were administered in-person by trained interviewers, 4-10 days apart. Trained nutrition professionals used Survey Net, matching foods consumed with 8-digit codes from the Food and Nutrient Database for Dietary Studies (FNDDS) version 3.0,(38) and My pyramid equivalents database for food groups (MPED 2: http://www.ars.usda.gov/SP2UserFiles/Place/80400530/pdf/mped/mped2_doc.pdf). Dietary vitamin D was among the nutrients made available by the FNDDS, from which daily values could be estimated and expressed in µg/d, using the average from the two 24-hr recalls conducted at baseline.

Supplemental vitamin D The HANDLS dietary supplement questionnaire was adapted from the 2007 NHANES instrument.(39) HANDLS participants provided supplement bottles during their dietary interview at the follow-up visit only (i.e. visit 2). Information on Over-The-Counter (OTC) vitamin and mineral supplements, antacids, prescription supplements, and botanicals were reported, and supplement users were asked about dose strength, dose amount consumed, length of supplement use (converted to days), frequency of use (daily, monthly, seasonally, annually), and if each supplement was taken the day prior to interview.

A HANDLS dietary supplement database was developed by trained nutritionists and registered dietitians. This database consisted of 4 files integrated to generate daily intake of each nutrient consumed by a dietary supplement user. [See detailed description at the HANDLS study website: https://handls.nih.gov/]. Vitamin D supplemental intake was ascertained for visit 1 if the daily amount (IU/d) was non-zero at visit 2 and the length of time for intake was greater or equal than the length of time (days) between the two visits, per individual. Thus, HANDLS participant was either 0: non-vitamin D containing supplement user at baseline or follow-up, 1: vitamin-D containing supplement user at baseline and during follow-up, 2: vitamin-D containing supplement user during follow-up only.

Covariates Covariates included age, sex, race (White vs. African American), marital status, educational attainment (<High School (HS); HS, >HS), poverty income ratio (PIR<125% for "poor"), measured body mass index (BMI, kg/m2), opiate, marijuana or cocaine use ("current" vs. "never or former"), smoking status ("current" vs. "never or former") and the Wide Range Achievement Test (WRAT) letter and word reading subtotal scores to measure literacy. (See Supplemental Method 1) To assess depressive symptoms with focus on affective, depressed mood, the 20-item CES-D was used. Baseline CES-D total score was included in the analysis as a potential confounder in the association between vitamin D exposures and cognitive change or baseline performance. (See Supplemental Method 1) The Healthy Eating Index (HEI-2010) total score, based on two 24-hr recalls administered at baseline, was used as a measure of overall dietary quality. See steps for calculating HEI-2010 at http://appliedresearch.cancer.gov/tools/hei/tools.html and http://handls.nih.gov/06Coll-dataDoc.html. Further, season of baseline MRV exam was used as proxy for sunshine exposure and was included as covariate in all models. Finally, self-reported history of type 2 diabetes, hypertension, cardiovascular disease (stroke, congestive heart failure, non-fatal myocardial infarction or atrial fibrillation) and dyslipidemia at first-visit were considered as covariates.(40) Statistical analysis Using Stata 15.0 (41) and accounting for sampling weights, population estimates of means and proportions were obtained. Means across stratifying variables (e.g. age/sex or race) were compared using svy:reg, relationship between categorical variables using svy:tab and design-based F-tests. Further, mixed-effects regression models with 11 continuous cognitive test score(s) as alternative outcomes were conducted. In these models the time variable was interacted with several covariates including the main exposure variables, namely VITDserum, VITDdiet and VITDsuppl. The models assume missingness at random with time points ranging between ~1.5-2.0 visits/person. (42) Predictive margins were estimated and plotted across TIME, stratifying by exposure group, from selected mixed-effects regression models, particularly those showing significant associations in the total population.

Moderating effect of sex and age groups was tested by adding interaction terms to separate multivariable mixed-effects regressions (3-way and 4-way interaction terms between Time, exposure, Age group and sex) and stratifying by sex and age group to examine relationships among the following groups: (1) Younger men, (2) Older men, (3) Younger women, (4) Older women, whenever at least one 4-way interaction was deemed statistically significant. Further, moderating effects by race were also examined using a similar approach [(1) Whites, (2) African-Americans] (Supplemental method 2), given the well-known higher prevalence of vitamin D deficiency among African-Americans compared with Whites and the differential rates of increases in vitamin D status recently shown by age, sex and race groups.(43) Variable time of follow-up is accounted for in the mixed-effects regression model as annual rate of change in the outcome was of primary interest.

Moreover, selection bias may occur due to non-random selection of participants with complete data from the target study population. Thus, in each mixed-effect regression model, a 2-stage Heckman selection process was conducted, by running a probit model to compute an inverse mills ratio at the first stage (derived from the predicted probability of being selected, conditional on the covariates in the probit model, mainly baseline age, sex, race, poverty status and education). At the second stage, this inverse mills ratio was then entered as a covariate in the final mixed-effects regression model, as was done in a previous study.(44) In all analyses, a type I error of 0.05 was considered for main effects whereas a p<0.10 was deemed significant for interaction terms,(45), prior to correcting for multiple testing. A familywise Bonferroni procedure was used to correct for multiple testing by accounting only for cognitive tests and assuming that exposures related to separate substantive hypotheses.(46) Therefore, for main effects, p<0.004 (0.05/11) was considered significant. Due to their lower statistical power compared to main effects, 2-way interaction terms had their critical p-values reduced to (0.10/11=0.009), while 3-way and 4-way interaction terms had their critical p-value reduced to 0.05. A similar approach was adopted in two other studies. (47, 48)

ELIGIBILITY:
Inclusion Criteria:

* HANDLS initially recruited 3,720 participants (Phase I, visit 1). Given that only Phase II had in-depth data including biochemical indices and cognitive performance measures, 25(OH)D was available for 1,981 participants at baseline. The corresponding sample size for dietary and supplemental vitamin D were N=2,177 and N=2,159, respectively. Complete and reliable cognitive tests at each visit varied in sample size as well. Further, the final analytic sample was determined based on exposure and covariate non-missingness at baseline and outcome non-missingness at either visit. The final analytic sizes ranged between N=1,231 and N=1,803 with k=1.5-1.9 observation/participant.

Exclusion Criteria:

* HANDLS participants with missing data on cognitive test score on both visits and/or missing data on exposure and covariates included in the mixed-effects regression models.

Ages: 30 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Serum 25(OH)D was lower among African-Americans who had a higher prevalence of vitamin D deficiency compared with Whites, in addition to consuming a smaller amount of vitamin D in the diet. Older participants tended to have a significant increase in serum 25(OH)D over time compared with younger men. Finally, older participants were more likely than younger men to be vitamin D-containing supplement users.
Sampling Method: Probability Sample
Enrollment: 3720 (Actual)
Dates: Start 2004-08-18 (Actual); Primary Completion 2013-07-07 (Actual); Study Completion 2013-07-07 (Actual)

PRIMARY OUTCOMES:
Cognitive change | Over a mean of 4.8 y
  Annual rate of change in cognitive test scores spanning several domains of cognition

CONTACTS AND LOCATIONS:
Locations (1):
- Biomedical Research Center, NIA/NIH/IRP, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzheimer's Association. 2009 Alzheimer's disease facts and figures. Alzheimers Dement. 2009 May;5(3):234-70. doi: 10.1016/j.jalz.2009.03.001. PMID 19426951
- [Background] Beydoun MA, Beydoun HA, Gamaldo AA, Teel A, Zonderman AB, Wang Y. Epidemiologic studies of modifiable factors associated with cognition and dementia: systematic review and meta-analysis. BMC Public Health. 2014 Jun 24;14:643. doi: 10.1186/1471-2458-14-643. PMID 24962204
- [Background] Buell JS, Dawson-Hughes B. Vitamin D and neurocognitive dysfunction: preventing "D"ecline? Mol Aspects Med. 2008 Dec;29(6):415-22. doi: 10.1016/j.mam.2008.05.001. Epub 2008 May 13. PMID 18579197
- [Background] McCann JC, Ames BN. Is there convincing biological or behavioral evidence linking vitamin D deficiency to brain dysfunction? FASEB J. 2008 Apr;22(4):982-1001. doi: 10.1096/fj.07-9326rev. Epub 2007 Dec 4. PMID 18056830
- [Background] Miller JW. Vitamin D and cognitive function in older adults: are we concerned about vitamin D-mentia? Neurology. 2010 Jan 5;74(1):13-5. doi: 10.1212/WNL.0b013e3181c719a2. Epub 2009 Nov 25. No abstract available. PMID 19940269
- [Background] Berridge MJ. Vitamin D cell signalling in health and disease. Biochem Biophys Res Commun. 2015 Apr 24;460(1):53-71. doi: 10.1016/j.bbrc.2015.01.008. PMID 25998734
- [Background] Eyles DW, Burne TH, McGrath JJ. Vitamin D, effects on brain development, adult brain function and the links between low levels of vitamin D and neuropsychiatric disease. Front Neuroendocrinol. 2013 Jan;34(1):47-64. doi: 10.1016/j.yfrne.2012.07.001. Epub 2012 Jul 11. PMID 22796576
- [Background] Etgen T, Sander D, Bickel H, Sander K, Forstl H. Vitamin D deficiency, cognitive impairment and dementia: a systematic review and meta-analysis. Dement Geriatr Cogn Disord. 2012;33(5):297-305. doi: 10.1159/000339702. Epub 2012 Jul 2. PMID 22759681
- [Background] Perna L, Mons U, Kliegel M, Brenner H. Serum 25-hydroxyvitamin D and cognitive decline: a longitudinal study among non-demented older adults. Dement Geriatr Cogn Disord. 2014;38(3-4):254-63. doi: 10.1159/000362870. Epub 2014 Jun 25. PMID 24969663
- [Background] Bartali B, Devore E, Grodstein F, Kang JH. Plasma vitamin D levels and cognitive function in aging women: the nurses' health study. J Nutr Health Aging. 2014 Apr;18(4):400-6. doi: 10.1007/s12603-013-0409-9. PMID 24676321
- [Background] Annweiler C, Rolland Y, Schott AM, Blain H, Vellas B, Beauchet O. Serum vitamin D deficiency as a predictor of incident non-Alzheimer dementias: a 7-year longitudinal study. Dement Geriatr Cogn Disord. 2011;32(4):273-8. doi: 10.1159/000334944. Epub 2012 Jan 19. PMID 22261995
- [Background] Annweiler C, Rolland Y, Schott AM, Blain H, Vellas B, Herrmann FR, Beauchet O. Higher vitamin D dietary intake is associated with lower risk of alzheimer's disease: a 7-year follow-up. J Gerontol A Biol Sci Med Sci. 2012 Nov;67(11):1205-11. doi: 10.1093/gerona/gls107. Epub 2012 Apr 13. PMID 22503994
- [Background] Llewellyn DJ, Lang IA, Langa KM, Muniz-Terrera G, Phillips CL, Cherubini A, Ferrucci L, Melzer D. Vitamin D and risk of cognitive decline in elderly persons. Arch Intern Med. 2010 Jul 12;170(13):1135-41. doi: 10.1001/archinternmed.2010.173. PMID 20625021
- [Background] Slinin Y, Paudel M, Taylor BC, Ishani A, Rossom R, Yaffe K, Blackwell T, Lui LY, Hochberg M, Ensrud KE; Study of Osteoporotic Fractures Research Group. Association between serum 25(OH) vitamin D and the risk of cognitive decline in older women. J Gerontol A Biol Sci Med Sci. 2012 Oct;67(10):1092-8. doi: 10.1093/gerona/gls075. Epub 2012 Mar 27. PMID 22454371
- [Background] Toffanello ED, Coin A, Perissinotto E, Zambon S, Sarti S, Veronese N, De Rui M, Bolzetta F, Corti MC, Crepaldi G, Manzato E, Sergi G. Vitamin D deficiency predicts cognitive decline in older men and women: The Pro.V.A. Study. Neurology. 2014 Dec 9;83(24):2292-8. doi: 10.1212/WNL.0000000000001080. Epub 2014 Nov 5. PMID 25378671
- [Background] Moon JH, Lim S, Han JW, Kim KM, Choi SH, Kim KW, Jang HC. Serum 25-hydroxyvitamin D level and the risk of mild cognitive impairment and dementia: the Korean Longitudinal Study on Health and Aging (KLoSHA). Clin Endocrinol (Oxf). 2015 Jul;83(1):36-42. doi: 10.1111/cen.12733. Epub 2015 Mar 4. PMID 25641087
- [Background] Miller JW, Harvey DJ, Beckett LA, Green R, Farias ST, Reed BR, Olichney JM, Mungas DM, DeCarli C. Vitamin D Status and Rates of Cognitive Decline in a Multiethnic Cohort of Older Adults. JAMA Neurol. 2015 Nov;72(11):1295-303. doi: 10.1001/jamaneurol.2015.2115. PMID 26366714
- [Background] Kuzma E, Soni M, Littlejohns TJ, Ranson JM, van Schoor NM, Deeg DJ, Comijs H, Chaves PH, Kestenbaum BR, Kuller LH, Lopez OL, Becker JT, Langa KM, Henley WE, Lang IA, Ukoumunne OC, Llewellyn DJ. Vitamin D and Memory Decline: Two Population-Based Prospective Studies. J Alzheimers Dis. 2016;50(4):1099-108. doi: 10.3233/JAD-150811. PMID 26836174
- [Background] Maddock J, Geoffroy MC, Power C, Hypponen E. 25-Hydroxyvitamin D and cognitive performance in mid-life. Br J Nutr. 2014 Mar 14;111(5):904-14. doi: 10.1017/S0007114513003176. Epub 2013 Oct 18. PMID 24135155
- [Background] Przybelski RJ, Binkley NC. Is vitamin D important for preserving cognition? A positive correlation of serum 25-hydroxyvitamin D concentration with cognitive function. Arch Biochem Biophys. 2007 Apr 15;460(2):202-5. doi: 10.1016/j.abb.2006.12.018. Epub 2007 Jan 8. PMID 17258168
- [Background] Buell JS, Scott TM, Dawson-Hughes B, Dallal GE, Rosenberg IH, Folstein MF, Tucker KL. Vitamin D is associated with cognitive function in elders receiving home health services. J Gerontol A Biol Sci Med Sci. 2009 Aug;64(8):888-95. doi: 10.1093/gerona/glp032. Epub 2009 Apr 17. PMID 19377013
- [Background] Lee DM, Tajar A, Ulubaev A, Pendleton N, O'Neill TW, O'Connor DB, Bartfai G, Boonen S, Bouillon R, Casanueva FF, Finn JD, Forti G, Giwercman A, Han TS, Huhtaniemi IT, Kula K, Lean ME, Punab M, Silman AJ, Vanderschueren D, Wu FC; EMAS study group. Association between 25-hydroxyvitamin D levels and cognitive performance in middle-aged and older European men. J Neurol Neurosurg Psychiatry. 2009 Jul;80(7):722-9. doi: 10.1136/jnnp.2008.165720. Epub 2009 May 21. PMID 19460797
- [Background] Llewellyn DJ, Langa KM, Lang IA. Serum 25-hydroxyvitamin D concentration and cognitive impairment. J Geriatr Psychiatry Neurol. 2009 Sep;22(3):188-95. doi: 10.1177/0891988708327888. Epub 2008 Dec 10. PMID 19073839
- [Background] Annweiler C, Schott AM, Rolland Y, Blain H, Herrmann FR, Beauchet O. Dietary intake of vitamin D and cognition in older women: a large population-based study. Neurology. 2010 Nov 16;75(20):1810-6. doi: 10.1212/WNL.0b013e3181fd6352. PMID 21079183
- [Background] Llewellyn DJ, Lang IA, Langa KM, Melzer D. Vitamin D and cognitive impairment in the elderly U.S. population. J Gerontol A Biol Sci Med Sci. 2011 Jan;66(1):59-65. doi: 10.1093/gerona/glq185. Epub 2010 Nov 1. PMID 21041201
- [Background] Breitling LP, Perna L, Muller H, Raum E, Kliegel M, Brenner H. Vitamin D and cognitive functioning in the elderly population in Germany. Exp Gerontol. 2012 Jan;47(1):122-7. doi: 10.1016/j.exger.2011.11.004. Epub 2011 Nov 21. PMID 22123431
- [Background] Andreeva VA, Whegang-Youdom S, Touvier M, Assmann KE, Fezeu L, Hercberg S, Galan P, Kesse-Guyot E. Midlife dietary vitamin D intake and subsequent performance in different cognitive domains. Ann Nutr Metab. 2014;65(1):81-9. doi: 10.1159/000365154. Epub 2014 Sep 16. PMID 25227981
- [Background] Chei CL, Raman P, Yin ZX, Shi XM, Zeng Y, Matchar DB. Vitamin D levels and cognition in elderly adults in China. J Am Geriatr Soc. 2014 Nov;62(11):2125-9. doi: 10.1111/jgs.13082. Epub 2014 Oct 3. PMID 25283584
- [Background] Assmann KE, Touvier M, Andreeva VA, Deschasaux M, Constans T, Hercberg S, Galan P, Kesse-Guyot E. Midlife plasma vitamin D concentrations and performance in different cognitive domains assessed 13 years later. Br J Nutr. 2015 May 28;113(10):1628-37. doi: 10.1017/S0007114515001051. Epub 2015 Apr 13. PMID 25864611
- [Background] Brouwer-Brolsma EM, Dhonukshe-Rutten RA, van Wijngaarden JP, van de Zwaluw NL, in 't Veld PH, Wins S, Swart KM, Enneman AW, Ham AC, van Dijk SC, van Schoor NM, van der Velde N, Uitterlinden AG, Lips P, Kessels RP, Steegenga WT, Feskens EJ, de Groot LC. Cognitive Performance: A Cross-Sectional Study on Serum Vitamin D and Its Interplay With Glucose Homeostasis in Dutch Older Adults. J Am Med Dir Assoc. 2015 Jul 1;16(7):621-7. doi: 10.1016/j.jamda.2015.02.013. Epub 2015 Mar 30. PMID 25838206
- [Background] Jorde R, Mathiesen EB, Rogne S, Wilsgaard T, Kjaergaard M, Grimnes G, Schirmer H. Vitamin D and cognitive function: The Tromso Study. J Neurol Sci. 2015 Aug 15;355(1-2):155-61. doi: 10.1016/j.jns.2015.06.009. Epub 2015 Jun 7. PMID 26092373
- [Background] Maddock J, Cavadino A, Power C, Hypponen E. 25-hydroxyvitamin D, APOE varepsilon4 genotype and cognitive function: findings from the 1958 British birth cohort. Eur J Clin Nutr. 2015 Apr;69(4):505-8. doi: 10.1038/ejcn.2014.201. Epub 2014 Oct 8. PMID 25293430
- [Background] Annweiler C, Milea D, Whitson HE, Cheng CY, Wong TY, Ikram MK, Lamoureux EL, Sabanayagam C. Vitamin D insufficiency and cognitive impairment in Asians: a multi-ethnic population-based study and meta-analysis. J Intern Med. 2016 Sep;280(3):300-11. doi: 10.1111/joim.12491. Epub 2016 Apr 1. PMID 27037788
- [Background] Nagel G, Herbolsheimer F, Riepe M, Nikolaus T, Denkinger MD, Peter R, Weinmayr G, Rothenbacher D, Koenig W, Ludolph AC, von Arnim CA; ActiFE Study group. Serum Vitamin D Concentrations and Cognitive Function in a Population-Based Study among Older Adults in South Germany. J Alzheimers Dis. 2015;45(4):1119-26. doi: 10.3233/JAD-143219. PMID 25649649
- [Background] Evans MK, Lepkowski JM, Powe NR, LaVeist T, Kuczmarski MF, Zonderman AB. Healthy aging in neighborhoods of diversity across the life span (HANDLS): overcoming barriers to implementing a longitudinal, epidemiologic, urban study of health, race, and socioeconomic status. Ethn Dis. 2010 Summer;20(3):267-75. PMID 20828101
- [Background] Powe CE, Evans MK, Wenger J, Zonderman AB, Berg AH, Nalls M, Tamez H, Zhang D, Bhan I, Karumanchi SA, Powe NR, Thadhani R. Vitamin D-binding protein and vitamin D status of black Americans and white Americans. N Engl J Med. 2013 Nov 21;369(21):1991-2000. doi: 10.1056/NEJMoa1306357. PMID 24256378
- [Background] Moshfegh AJ, Rhodes DG, Baer DJ, Murayi T, Clemens JC, Rumpler WV, Paul DR, Sebastian RS, Kuczynski KJ, Ingwersen LA, Staples RC, Cleveland LE. The US Department of Agriculture Automated Multiple-Pass Method reduces bias in the collection of energy intakes. Am J Clin Nutr. 2008 Aug;88(2):324-32. doi: 10.1093/ajcn/88.2.324. PMID 18689367
- [Background] Beydoun MA, Tajuddin SM, Dore GA, Canas JA, Beydoun HA, Evans MK, Zonderman AB. Vitamin D Receptor and Megalin Gene Polymorphisms Are Associated with Longitudinal Cognitive Change among African-American Urban Adults. J Nutr. 2017 Jun;147(6):1048-1062. doi: 10.3945/jn.116.244962. Epub 2017 Apr 26. PMID 28446629
- [Background] Ibrahim JG, Molenberghs G. Missing data methods in longitudinal studies: a review. Test (Madr). 2009 May 1;18(1):1-43. doi: 10.1007/s11749-009-0138-x. PMID 21218187
- [Background] Schleicher RL, Sternberg MR, Lacher DA, Sempos CT, Looker AC, Durazo-Arvizu RA, Yetley EA, Chaudhary-Webb M, Maw KL, Pfeiffer CM, Johnson CL. The vitamin D status of the US population from 1988 to 2010 using standardized serum concentrations of 25-hydroxyvitamin D shows recent modest increases. Am J Clin Nutr. 2016 Aug;104(2):454-61. doi: 10.3945/ajcn.115.127985. Epub 2016 Jul 6. PMID 27385610
- [Background] Beydoun MA, Beydoun HA, Kitner-Triolo MH, Kaufman JS, Evans MK, Zonderman AB. Thyroid hormones are associated with cognitive function: moderation by sex, race, and depressive symptoms. J Clin Endocrinol Metab. 2013 Aug;98(8):3470-81. doi: 10.1210/jc.2013-1813. Epub 2013 May 20. PMID 23690311
- [Background] Beydoun MA, Beydoun HA, Rostant OS, Dore GA, Fanelli-Kuczmarski MT, Evans MK, Zonderman AB. Thyroid hormones are associated with longitudinal cognitive change in an urban adult population. Neurobiol Aging. 2015 Nov;36(11):3056-3066. doi: 10.1016/j.neurobiolaging.2015.08.002. Epub 2015 Aug 8. PMID 26329688
- [Background] Beydoun MA, Canas JA, Dore GA, Beydoun HA, Rostant OS, Fanelli-Kuczmarski MT, Evans MK, Zonderman AB. Serum Uric Acid and Its Association with Longitudinal Cognitive Change Among Urban Adults. J Alzheimers Dis. 2016 Apr 21;52(4):1415-30. doi: 10.3233/JAD-160028. PMID 27104899
- See also: S Department of Agriculture ARS, Food Surveys Research Group. USDA Food and Nutrient Database for Dietary Studies, 3.0 — http://www.ars.usda.gov/Services/docs.htm?docid=12089.
- See also: Centers for Disease Control and Prevention — https://wwwn.cdc.gov/nchs/nhanes/continuousnhanes/default.aspx?BeginYear=2007
- See also: STATA. Statistics/Data Analysis: Release 15.0. Texas: Stata Corporation, 2017 — http://www.stata.com
- See also: Selvin S. Statistical Analysis of Epidemiologic Data. 3rd ed: Oxford University Press, 2004. — https://books.google.com/books/about/Statistical_Analysis_of_Epidemiologic_Da.html?id=EpEfWvk8mS4C
- See also: Hochberg Y, Tamhane, A. C.,. Multiple comparison procedures. New York: Wiley, 1987. — https://books.google.com/books?id=qxnvAAAAMAAJ&q=Multiple+comparison+procedures&dq=Multiple+comparison+procedures&hl=en&sa=X&ved=0ahUKEwj96siun4DXAhUoqVQKHUwzAtgQ6AEINTAC